CLINICAL TRIAL: NCT00591435
Title: Resident Training Affects Intra-Operative Workflow and Costs
Brief Title: Influence of Resident Training on Intra-operative Workflow
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: Department of Anaesthesiology and Intensive Care Medicine (Ambiguous)
Responsible Party: Jens Scholz, Professor of Anaesthesiology, Chair of the Department of Anaesthesiology and Intensive Care Medicine
Other Study IDs: UKSH_Hanss; IRB: A138/07
Record Dates: First submitted 2007-12-28; First posted 2008-01-11 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2007-11

CONDITIONS: Intraoperative Workflow; Anesthesia and Procedure Related Time Intervals
Keywords: Anesthesia; Surgery; Education; Economics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: 200 laparoscopic cholecystectomies will be included, consultant cases will be compared to resident cases
  Interventions: Other: Comparison of performance of consultants versus residents
- 2: 200 laparoscopic pelviscopies will be included, consultant cases will be compared to resident cases
  Interventions: Other: Comparison of performance of consultants versus residents
- 3: 200 transurethral resection of urinary bladder or prostate gland will be included, consultant cases will be compared to resident cases
  Interventions: Other: Comparison of performance of consultants versus residents

INTERVENTIONS:
Other: Comparison of performance of consultants versus residents — Anesthesia as well as surgical workflow will be analysed. Performance of consultants will be compared to residents

SUMMARY:
Anaesthesia and surgery related time intervals of three standard operations are compared depending on whether residents or consultants are performing anaesthesia and surgery.

Hypothesis: Perioperative workflow is influenced by state of education, time intervals reflecting anaesthesia as well as surgical performance increase due to resident training. Therefore, costs of perioperative care increase as well.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects scheduled for one of the three defined procedures (defined by German Diagnose Related Groups ID) under general or regional anesthesia

Exclusion Criteria:

* Patient's refusal of data collection, emergency procedures, change of physician in charge (resident to consultant or the other way around) of anesthesia or surgical team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy subjects scheduled for one of the three defined procedures (defined by German Diagnose Related Groups ID) under general or regional anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2007-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Anaesthesia and procedural related time intervals | All events will be recorded intraoperativly

SECONDARY OUTCOMES:
OR costs are calculated as $ 15.00 per minute, additional costs due to increase of time intervals will be analyzed | All data will be recorded intraoperaitvly

CONTACTS AND LOCATIONS:
Overall Officials: Jens Scholz, MD, Professor, Principal Investigator — Department of Anaesthesiology and Intenisve Care Medicine, University Hospital Schleswig-Holstein, Campus Kiel
Locations (1):
- University Hospital Schleswig-Holstein, Campus Kiel, Kiel, Schleswig-Holstein, Germany